CLINICAL TRIAL: NCT06487520
Title: The Effect of Different Images Watched Wiht Virtual Reality on Perception of Pain And Anxiety During Flebotomy
Brief Title: The Effect of Different Images Watched With Virtual Reality During Phlebotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Dilek Karaman, Associate Professor, Zonguldak Bulent Ecevit University, Ahmet Erdogan Health Services Vocational School, Health Care Services Program, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/04-18
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Pain Management; Anxiety Management; Blood Donation; Virtual Reality
Keywords: Pain; Anxiety; Phlebotomy; Blood Donation; Virtual Reality
MeSH Terms: conditions — Agnosia; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group watching hot environment image (Experimental): A virtual reality headset was placed on the heads of the individuals included in the intervention group one minute before the procedure and a cold environment image called "Peaceful mountain snow" was shown. By starting the image before the procedure, the individual was prevented from seeing the needle and blood. At the end of the procedure, the tourniquet and needle were removed and the virtual reality headset was removed from the individual's head and the displayed image was terminated.
  Interventions: Other: group watching hot environment image
- group watching cold environment image (Placebo Comparator): A virtual reality headset was placed on the heads of the individuals in the placebo group one minute before the procedure and a warm environment image called "Deep space relaxation" was shown. By starting the image before the procedure, the individual was prevented from seeing the needle and blood. At the end of the procedure, the tourniquet and needle were removed and the virtual reality headset was removed from the individual's head and the image shown was terminated
  Interventions: Other: group watching cold environment image
- The control group (No Intervention): No intervention was performed on the control group before the peripheral intravenous catheterization procedure, and the standard peripheral intravenous catheterization procedure was performed.

INTERVENTIONS:
Other: group watching hot environment image — In this study, Sony playstation VR (Virtual Reality) glasses with LCD (Liquid Crystal Display) screen with OLED (Organic Light-Emitting Diode) technology and 1080P resolution integrated on the device were used. These glasses work integrated with the processor box. The processor box, which provides communication with the Sony playstation VR glasses, can also be connected to the computer with HDMI (High Definition Multimedia Interface) output. Within the scope of the study, the licensed "Peaceful mountain snow" image was shown. This image includes a cold winter day.
  Following the completion of every VR session, the removable face pad was replaced and the goggles and headsets were wiped down with alcohol-based sanitary wipes. Preventing infection via the sharing of the technology was a paramount issue with the study patients.
  Arms: group watching hot environment image
Other: group watching cold environment image — In this study, Sony playstation VR (Virtual Reality) glasses with LCD (Liquid Crystal Display) screen with OLED (Organic Light-Emitting Diode) technology and 1080P resolution integrated on the device were used. These glasses work integrated with the processor box. The processor box, which provides communication with the Sony playstation VR glasses, can also be connected to the computer with HDMI (High Definition Multimedia Interface) output. Within the scope of the study, the licensed "Deep space relaxation" image was shown. This image contains a hot environment image with explosions in space.Following the completion of every VR session, the removable face pad was replaced and the goggles and headsets were wiped down with alcohol-based sanitary wipes. Preventing infection via the sharing of the technology was a paramount issue with the study patients.
  Arms: group watching cold environment image

SUMMARY:
Aim: The purpose of this study was to investigate the effect of watching a cold environment image via virtual reality on pain and anxiety related to phlebotomy procedure in volunteer blood donors.

Methods: The study was conducted between June 2019 and December 2019 with 120 healthy individuals who applied for blood donation for the first time in Northern Turkey. Individuals included in the study were assigned to intervention, placebo and control groups with 40 people in each group by block randomization method. During the phlebotomy procedure, the intervention group watched a cold environment image via virtual reality, the placebo group watched a hot environment image, and the control group received standard application. "Descriptive Characteristics Form", "Visual Comparison Scale", "State and Trait Anxiety Inventory" and The CONSORT checklist were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Being in accordance with time and place
* Being aged between 18 and 35 years
* Being able to evaluate the visual analog scale correctly
* Participating voluntarily in the research.
* Being willing to donate blood
* Donating blood for the first time
* Have a body mass index within normal limits (18.5-24.9 kg/m2)
* Have no vision or hearing problems
* Have no disease that may affect pain perception
* Have no vertigo, heart or lung disease
* Have no signs of infection, dermatitis, phlebitis, scar tissue or incision in the area where invasive intervention will be performed
* Have no psychiatric disease
* Being able to accurately assess the state and trait anxiety inventory with the VAS
* Have an average pressure pain threshold value of 8-16 Lb obtained from three measurements taken at 5-second intervals from the elbow region of the left upper extremity where no intervention was performed
* Have no vertigo, heart or lung disease
* Have no signs of infection, dermatitis, phlebitis, scar tissue or incision in the area where invasive intervention will be performed
* Have no psychiatric disease
* Being able to accurately assess the state and trait anxiety inventory with the VAS
* Have an average pressure pain threshold value of 8-16 pounds (Lb) obtained from three measurements taken at 5-second intervals from the elbow region of the left upper extremity where no intervention was performed

Exclusion Criteria:

* Not participating voluntarily in the research
* Not fitting the inclusion criteria of the research
* Having a vision or hearing problem
* Failure of phlebotomy at the first attempt
* Development of syncope after phlebotomy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
pain intensity in cm | 6 months
  The VAS is a 100 mm (10 cm) ruler that can be used horizontally or vertically. The value of "0" at the starting level defines painlessness, and the value of "10" at the ending level defines the most severe pain. The individual marks the intensity of pain they experience on this scale. In this study, the score measurements were determined in centimeters (cm) on the VAS prepared vertically to determine the intensity of pain experienced by individuals during phlebotomy application.individuals.during the procedure. One end indicated lack of pain and the other the most.Pain intensity was evaluated in centimeters.severe pain possible. Pain severity was evaluated in millimeters.
State-Trait Anxiety Inventory (STAI) score | 6 months
  The inventory is in the form of a 4-point Likert scale, and the items in the State and Trait Anxiety Subscales are marked according to the degree of severity of the emotions and behaviors. There are ten items in the State Anxiety Scale and seven items in the Trait Anxiety Scale that contain reversed statements.

SECONDARY OUTCOMES:
weight in kilograms | 6 months
  Body mass index normal weight (18.5-24.9 kg/m2)
Pressure pain threshold | 6 months
  The average value of the pressure pain threshold, which is defined as the point of pain.from three measurements taken at 5-second intervals from the elbow region of the left upper extremity where no intervention was performedperception and can vary from person to person, is between 8-16 Lb

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided